CLINICAL TRIAL: NCT01451086
Title: Safety and Immunogenicity of 23-valent Pneumococcal Polysaccharide Vaccine in 2 to 70 Years Old Healthy People in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20080808
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Safety; Immunogenicity; Pneumococcal vaccine
MeSH Terms: interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vaccine made by Beijing Minhai Biotechnology Co., Ltd (Experimental): Subjects receive 0.5 mL/dose of 23-valent pneumococcal polysaccharide vaccine by intramuscular (deltoid) injection on Day 0.
  Interventions: Biological: vaccine made by Beijing Minhai Biotechnology Co., Ltd
- vaccine made by Chengdu Institute of Biological Products (Active Comparator): Subjects receive 0.5 mL/dose of 23-valent pneumococcal polysaccharide vaccine by intramuscular (deltoid) injection on Day 0.
  Interventions: Biological: vaccine made by Chengdu Institute of Biological Products

INTERVENTIONS:
Biological: vaccine made by Beijing Minhai Biotechnology Co., Ltd — Subjects receive 0.5 mL/dose of 23-valent pneumococcal polysaccharide vaccine by intramuscular (deltoid) injection on Day 0.
  Arms: vaccine made by Beijing Minhai Biotechnology Co., Ltd
Biological: vaccine made by Chengdu Institute of Biological Products — Subjects receive 0.5 mL/dose of 23-valent pneumococcal polysaccharide vaccine by intramuscular (deltoid) injection on Day 0.
  Arms: vaccine made by Chengdu Institute of Biological Products

SUMMARY:
Pneumococcal infection is a leading cause of death throughout the world and a major cause of pneumonia, bacteremia, meningitis, and otitis media.

It has been established that purified pneumococcal capsular polysaccharides induce antibody production and such antibody is effective in preventing pneumococcal disease. Clinical studies have demonstrated the immunogenicity of each of the 23 capsular types when tested in polyvalent vaccines. Studies of 23-valent pneumococcal vaccine in children of two years old and older and in adults of all ages have showed immunogenic response. In order to provide more evidence for the immunogenicity and the safety of the vaccine, a phase III clinical trial is planed to conduct.

DETAILED DESCRIPTION:
Pneumonia is a major cause of morbidity and mortality in developing countries. Pneumonia is predominantly bacterial in origin: isolation rates of Streptococcus pneumoniae and Haemophilus influenzae were 34% and 40%, respectively, in a series of lung aspirates collected from children under 5 years of age (Shann et al., 1984).

Pneumococcal infection is a leading cause of death throughout the world and a major cause of pneumonia, bacteremia, meningitis, and otitis media.

Strains of drug-resistant S. pneumoniae have become increasingly common in China and in other parts of the world. In some areas as many as 35% of pneumococcal isolates have been reported to be resistant to penicillin. Many penicillin-resistant pneumococci are also resistant to other antimicrobial drugs (e.g., erythromycin, trimethoprim-sulfamethoxazole and extended-spectrum cephalosporins), therefore the importance of vaccine prophylaxis should be emphasized against pneumococcal disease.

Epidemiology Pneumococcal infection causes approximately125,000 deaths annually in China. At least 2,500,000 cases of pneumococcal pneumonia are estimated to occur annually in the United States; S. pneumoniae accounts for approximately 25-35% of cases of community-acquired bacterial pneumonia in persons who require hospitalization.

Despite appropriate antimicrobial therapy and intensive medical care, the overall case-fatality rate for pneumococcal bacteremia is 15-20% among adults, and among elderly patients this rate is approximately 30-40%. An overall case-fatality rate of 36% was documented for adult inner-city residents who were hospitalized for pneumococcal bacteremia.

Invasive pneumococcal disease (e.g., bacteremia or meningitis) and pneumonia cause high morbidity and mortality in spite of effective antimicrobial control by antibiotics. These effects of pneumococcal disease appear due to irreversible physiologic damage caused by the bacteria during the first 5 days following onset of illness, and occur regardless of antimicrobial therapy. Vaccination offers an effective mean of further reducing the mortality and morbidity of this disease.

Risk Factors In addition to the very young and persons 65 years of age or older, patients with certain chronic conditions are at increased risk of developing pneumococcal infection and severe pneumococcal illness.

Patients with chronic cardiovascular diseases (e.g., congestive heart failure or cardiomyopathy), chronic pulmonary diseases (e.g., chronic obstructive pulmonary disease or emphysema), or chronic liver diseases (e.g., cirrhosis), diabetes mellitus, alcoholism or asthma (when it occurs with chronic bronchitis, emphysema, or long-term use of systemic corticosteroids) have an increased risk of pneumococcal disease. In adults, this population is generally immunocompetent.

Patients at high risk are those who have a decreased responsiveness to polysaccharide antigen or an increased rate of decline in serum antibody concentration as a result of: immunosuppressive conditions (congenital immunodeficiency, human immunodeficiency virus (HIV) infection, leukemia, lymphoma, multiple myeloma, Hodgkin's disease, or generalized malignancy); organ or bone marrow transplantation; therapy with alkylating agents, antimetabolites, or systemic corticosteroids; chronic renal failure or nephrotic syndrome.

Patients at the highest risk of pneumococcal infection are those with functional or anatomic asplenia (e.g., sickle cell disease or splenectomy), because this condition leads to reduced clearance of encapsulated bacteria from the bloodstream. Children who have sickle cell disease or have had a splenectomy are at increased risk of outbreak pneumococcal sepsis associated with high mortality.

Immunogenicity It has been established that purified pneumococcal capsular polysaccharides induce antibody production and that such antibody is effective in preventing pneumococcal disease. Clinical studies have demonstrated the immunogenicity of each of the 23 capsular types when tested in polyvalent vaccines.

Studies of 23-valent pneumococcal vaccines in children of two years old and older and in adults of all ages have showed immunogenic responses. Protective capsular type-specific antibody levels generally develop in the third week following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 70 years on the day of inclusion
* Informed consent form signed by subjects and parent/guardian
* Subjects and parents/guardians able to attend all scheduled visits and comply with all study procedures

Exclusion Criteria:

* Subjects with any pneumococcal vaccine before vaccination
* History of pneumococcal infection
* Women in pregnancy or lactation period in trial period
* Allergic history or any SAE after vaccination, such as allergy, urticaria, dyspnea, angioedema, celialgia
* Known or suspected immune dysfunction, including persons with congenital immunodeficiency or persons with HIV positive.
* Functional or anatomic asplenia
* Patients treated with chemotherapy in past 5 years or administered with immunosuppressive agents, cytotoxicity factor or corticosteroids in the 6 months preceding the vaccine trial
* Receipt of blood or blood-derived products in the 3 months preceding vaccination
* Participation in another clinical study investigating a vaccine, drug in the 30 days preceding vaccination
* Receipt of any live virus vaccine in the 30 days preceding vaccination
* Receipt of any subunit vaccine and inactivated vaccine in the 14 days before vaccination
* Thrombocytopenia, bleeding disorder
* History of asthma，angioneurotic edema，diabetes mellitus or malignancy tumor
* History of thyroid gland excision or treatment for thyroid gland disease in last 12 months
* Hypertension, blood pressure still above 145/95mmHg even with drug treatment
* History of eclampsia, epilepsia, psychosis
* Febrile illness (temperature ≥ 38°C) in the 3 days or any acute illness/infection in the 7 days preceding vaccination
* In progress of anti-tuberculosis prophylaxis or therapy
* Those can not fulfill the protocol or can not sign the informed consent form for any medical, psychological, social, occupational and other reasons, according to investigator judgment

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of 23-valent Pneumococcal Polysaccharide Vaccine after vaccination | 28 days after vaccination
  To evaluate the percentage of subjects exhibiting a ≥ 2 fold increase in IGG antibody level after vaccination

SECONDARY OUTCOMES:
To evaluate the safety of 23-valent Pneumococcal Polysaccharide Vaccine after vaccination | 28 days after vaccination
  To evaluate the frequency of systemic and local adverse reactions in healthy subjects after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China